CLINICAL TRIAL: NCT04382625
Title: Hydroxychloroquine in SARS-CoV-2 (COVID-19) Pneumonia Trial
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: Secondary to other study results, suspended for a scientific review
Sponsor: Kootenai Health (Other)
Collaborators: Washington State University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 18244
Record Dates: First submitted 2020-04-14; First posted 2020-05-11 (Actual); Last update posted 2021-02-05 (Actual); Status verified 2020-05

CONDITIONS: SARS-CoV-2 Pneumonia; COVID-19
Keywords: SARS-CoV-2; Pneumonia; Hydroxychloroquine; COVID-19
MeSH Terms: conditions — COVID-19; Pneumonia | interventions — Hydroxychloroquine

STUDY DESIGN:
Intervention Model Description: Single-center pragmatic randomized open-label trial of hydroxychloroquine + usual care in hospitalized adults with confirmed SARS-CoV-2 infection and acute hypoxia compared to usual care.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Hydroxychloroquine (HCQ) (Experimental): Initial dose: HCQ 400mg x 2 (800mg) then 200mg by mouth, three times per day (600mg/24hr period) starting 8 hours after the initial dose for a total of 14 doses over 5 days Plus Usual Care (See below for full description)
  Interventions: Drug: Hydroxychloroquine
- Usual Care (No Intervention): The care of hospitalized patients with covid-19 is evolving with hospital guidelines arising across the U.S. with several commonalities. Patients receive clinical assessment, chest x-ray, covid-19 testing, basic labs (WBC, CMP), and additional labs based on protocol or clinical judgment (ABG, CRP, LDH), antibiotics for possible bacterial pneumonia, acetaminophen for fever, supplemental O2, and consideration for mechanical ventilation. Early intubation over escalating noninvasive support. Low tidal volume ventilation and prone positioning are lung protective strategies used in critically ill covid-19 patients that are based on management of acute respiratory distress syndrome generally. Conservative fluid replacement is used to avoid worsening oxygenation.

INTERVENTIONS:
Drug: Hydroxychloroquine — Hydroxychloroquine is currently widely used for treatment of autoimmune disease including systemic lupus erythematosus and rheumatoid arthritis, and it has been used to prevent and treat malaria.
  Other Names: Plaquenil
  Arms: Hydroxychloroquine (HCQ)

SUMMARY:
Novel coronavirus SARS(Severe Acute Respiratory Syndrome)-CoV-2 was first identified during the outbreak in Wuhan, China in December 2019 with the now resulting pandemic. Aggressive supportive care is the mainstay of treatment currently and rescue with lung protective mechanical ventilation is essential for survival in patients with severe acute respiratory distress syndrome. Despite supportive care, mortality is significant in hospitalized patients in the U.S., especially among patients > 65 years of age. Pharmacologic treatments to decrease disease severity are urgently needed. Hydroxychloroquine is currently widely used for treatment of autoimmune disease including systemic lupus erythematosus and rheumatoid arthritis, and it has been used to prevent and treat malaria. In vitro and in vivo antiviral activity towards SARS-CoV-2 has been reported. Since hydroxychloroquine has been used for decades its properties as a drug are well known. The investigators propose a pragmatic trial of hydroxychloroquine in moderately ill hospitalized adults with SARS-CoV-2 pneumonia with the hypothesis that hydroxychloroquine reduces severity of acute lung injury caused by SARS-CoV-2 infection.

DETAILED DESCRIPTION:
Novel coronavirus SARS-CoV-2 was first identified during the outbreak in Wuhan, China in December 2019 with the now resulting pandemic. Aggressive supportive care is the mainstay of treatment currently and rescue with lung protective mechanical ventilation is essential for survival in patients with severe acute respiratory distress syndrome. Despite supportive care, mortality is significant in hospitalized patients in the U.S., especially among patients > 65 years of age. Pharmacologic treatments to decrease disease severity are urgently needed. Candidate treatments with antiviral activity and/or immune-modulating effects include hydroxychloroquine (HCQ), lopinavir/ritonavir, remdesivir, and tocilizumab among others. There is limited high quality clinical data prompting a dilemma of how to use and review potential treatments and ensure patient safety now as the pandemic begins to peak. There are also significant limitations in drug supplies at many institutions.

Hydroxychloroquine is currently widely used for treatment of autoimmune disease including systemic lupus erythematosus and rheumatoid arthritis, and it has been used to prevent and treat malaria. In vitro and in vivo antiviral activity towards SARS-CoV-2 has been reported. Since hydroxychloroquine has been used for decades its properties as a drug are well known. Pertinent adverse events to monitor in a hospitalized patient include QTc (corrected QT interval) prolongation, elevation of liver enzymes/acute liver injury, and hypokalemia.

Acute lung injury and progressive respiratory failure is the major cause of mortality in SARS-CoV-2 infection. In acute lung injury and respiratory distress syndrome, the severity of hypoxia is categorized by the Pao2/FIO2 (fraction of inspired oxygen) ration as mild (200 mm Hg<Pao2/Fio2≤300 mm Hg), moderate (100 mm Hg<Pao2/Fio2≤200 mm Hg), and severe (Pao2/Fio2 ≤100 mm Hg). A persistently low Pao2/Fio2 ratio is associated with worse outcomes and may be a marker of failure to respond to conventional therapy. PaO2/FIO2 is a clinically useful measure in patients regardless of if they are receiving noninvasive supplemental O2 or mechanical ventilation, and low ratios are associated with duration of ICU stay and hospital mortality.

The care of hospitalized patients with covid-19 is evolving with hospital guidelines arising across the U.S. with several commonalities. Patients receive clinical assessment, chest x-ray, covid-19 testing, basic labs (WBC, CMP), and additional labs based on protocol or clinical judgment (ABG, CRP-C reactive protein, LDH), antibiotics for possible bacterial pneumonia, acetaminophen for fever, supplemental O2, close monitoring for worsening respiratory status and consideration for mechanical ventilation. Since covid-19 is a novel illness, there is no proven clinically efficacious drug treatment. Candidate drugs are being used, some in the context of trials and others by physician discretion. Early intubation over escalating noninvasive support (ie. High flow nasal canula and bipap) has been adopted due to the frequency of rapidly worsening oxygenation, hemodynamic instability, and to protect staff from virus aerosolization. Low tidal volume ventilation and prone positioning are lung protective strategies used in critically ill covid-19 patients that are based on management of acute respiratory distress syndrome generally. Arrhythmias, cardiomyopathy, and shock are serious complications from covid-19 that warrant avoidance of acidosis, electrolyte monitoring and replacement, and pressor support. Conservative fluid replacement is used to avoid worsening oxygenation. In sum, multiple factors including timeliness and quality of care likely affect patient outcomes. Hospitalists and pulmonary critical care physicians direct the care of covid-19 patients with support from specialists as needed including infectious disease, cardiology, and nephrology.

Pragmatic trials focus on studying the real-world effect of an intervention, such as a medication, in the context of other care a patient is likely to receive. The intervention is delivered by staff normally taking care of the patient with monitoring that is routinely available. Advantages can include generalizability, increased physician participation due to less burdensome study protocols, and feasibility. Disadvantages include allowance of unblinded design, bias from physicians and patients about the intervention, and more heterogeneity in treatment than in a mechanistic protocolized trial. Efforts to minimize bias include selecting objective outcomes (e.g. PaO2/FIO2 rather than cough or dyspnea).

ELIGIBILITY:
Inclusion Criteria:

1. Age > 18 years of age
2. SARS-CoV-2 positive per FDA approved RT-PCR (reverse transcription-polymerase chain reaction)
3. Acute hypoxia (O2 sat < 90 % or paO2 < 60 on room air), or above baseline chronic O2 requirement
4. Inpatient admission

Exclusion Criteria:

1. Requires supplemental O2 >10 litres per minute or mechanical ventilation on admission
2. Pregnancy
3. AST/ALT > 5 times the upper limit normal
4. Baseline prolonged QT
5. Child-Pugh Score B or greater
6. ESRD(end-stage renal disease) requiring dialysis
7. Known allergy to medication component,
8. History of severe G6PD (glucose-6-phosphate dehydrogenase)
9. Myasthenia gravis
10. Porphyria
11. Ongoing treatment for epilepsy
12. Life expectancy < 6 months,
13. Patient lacks capacity to provide consent and does not have a surrogate decision maker.
14. Retinal Disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-10 (Estimated); Primary Completion 2022-01-01 (Estimated); Study Completion 2022-06-01 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline Oxygenation on Day 1 to Day 5 | Day 1 of treatment to day 5 of treatment
  paO2
Change from Baseline Oxygenation at Day 5 | Day 1 of treatment to day 5 of treatment
  FIO2

SECONDARY OUTCOMES:
Intensive Care length of stay | Day 0 to Day 28
  Length in hours
Required Mechanical Ventilation | Day 0 to Day 28
  Length in hours
Required Oxygen supplementation | Day 0 to Day 28
  Length in hours
Hospitalization length of Stay | Day 0 to Day 28
  Length in hours
Mortality | Day 0 to Day 28
  Date of Death
Cardiac Arrhythmia - Polymorphic Ventricular Tachycardia | Day 0 to Day 28
  Cardiologist Diagnostic Documentation
Cardiac Arrhythmia - Ventricular Tachycardia | Day 0 to Day 28
  Cardiologist Diagnostic Documentation
Cardiac Arrhythmia - Lengthening QTc | Day 0 to Day 28
  Cardiologist Diagnostic Documentation

CONTACTS AND LOCATIONS:
Overall Officials: Sean Cook, D.O., Principal Investigator — Kootenai Health; Jeanette Berg, MD, PhD, Principal Investigator — Kootenai Health; Sterling McPherson, PhD, Principal Investigator — Washington State University; John Roll, PhD, Principal Investigator — Washington State University
Locations (1):
- Kootenai Health, Coeur d'Alene, Idaho, United States

IPD SHARING:
Plan to Share IPD: No